CLINICAL TRIAL: NCT05018416
Title: A Phase 2, Randomized, Open-Labeled, Repeat Dose, Safety and Efficacy Study of Renal Autologous Cell Therapy (REACT) in Subjects With Type 1 or 2 Diabetes and Chronic Kidney Disease (REGEN-007)
Brief Title: Study of Renal Autologous Cell Therapy (REACT) in Subjects With Type 1 or 2 Diabetes and Chronic Kidney Disease (REGEN-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REGEN-007
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Kidney Biopsy; REACT
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 REACT injections (Experimental): Cohort 1 subjects will receive 2 REACT injections in the biopsied and non-biopsied contralateral kidneys 3 months apart (+60 days).
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)
- 1 REACT Injection (Experimental): Cohort 2 subjects will receive 1 REACT injection into the biopsied kidney and if a pre-defined trigger is met, will undergo a second REACT injection into the contralateral kidney.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Autologous selected renal cells (SRC)

SUMMARY:
The purpose of this study is to assess the safety, efficacy, and durability of up to two REACT injections delivered percutaneously into biopsied and non-biopsied contralateral kidneys on renal function progression in two different cohorts of subjects with T1DM or T2DM and CKD.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety, efficacy, and durability of up to two REACT injections delivered percutaneously into biopsied and non-biopsied contralateral kidneys on renal function progression in two different cohorts of subjects with T1DM or T2DM and CKD:

* Cohort 1: Two scheduled REACT injections given 3 months (+60 days) with at least 18- month follow-up
* Cohort 2: One scheduled REACT injection with a possible second REACT injection, no less than 3 months after the first one, within 30 days (+30 days) of meeting a renal function redose trigger (triggered up to 15 months following the first REACT injection).

Both cohorts will be followed for 18 months after the final REACT injection. If a Cohort 2 subject does not meet a trigger, the subject will be followed for at least 18 months after the first injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 30 to 80 years, inclusive, on the date informed consent is signed.
2. Clinical diagnosis of T1DM or T2DM, controlled per institutional standard of care.
3. The subject has a clinical diagnosis of diabetic nephropathy as the underlying cause of renal disease (diagnosis does not have to be confirmed via renal biopsy).
4. The subject has a serum glycosylated hemoglobin (HbA1c) level less than 10% at the Screening Visit.
5. The subject has a documented clinical diagnosis of an eGFR between 20 and 50 mL/min/1.73m² inclusive not requiring renal dialysis.

Exclusion Criteria:

1. The subject has a history of renal transplantation.
2. The subject has a mean systolic blood pressure greater than or equal to 140 mmHg and/or mean diastolic blood pressure greater than or equal to 90 mmHg at screening.

   Subjects with blood pressure outside of this range prior to biopsy/injection may continue if approved by the Medical Monitor.
3. The subject has hemoglobin levels less than 10 g/dL and is not responsive to the standard medical intervention for CKD-related anemia prior to randomization.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Improvement in renal function progression rate as indicated by the change from pre-injection baseline value in total (acute + chronic) slope of estimated glomerular filtration rate (eGFR) using the CKD-EPI 2009 equation | Screening thru month 28
Procedural and investigational product-related treatment-emergent adverse events (TEAEs) obtained through 18 months after the last REACT injection. | Screening thru 18 months after the last injection of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Taylor, Study Director — Prokidney
Locations (5):
- United States (5):
  - Kidney Associates of Colorado, P.C. - Frenova, Denver, Colorado
  - Nephrology Associates, Newark, Delaware
  - Boise Kidney and Hypertension Institute - Frenova, Nampa, Idaho
  - Paragon Health, PC d/b/a Nephrology Center, PC - Frenova, Kalamazoo, Michigan
  - Nephrology and Hypertension Associates Ltd - Frenova, Tupelo, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cizman B, Butler EL, Stavas J, Prakash R, Saad T, Silva A, Wooldridge T, Aqeel A, Yan H, Barysauskas CM, Culleton B. A Randomized Clinical Trial of Kidney Autologous Cell Therapy in Diabetic Kidney Disease. Clin J Am Soc Nephrol. 2026 Jan 2. doi: 10.2215/CJN.0000000969. Online ahead of print. No abstract available. PMID 41481370